CLINICAL TRIAL: NCT02667275
Title: A Randomized, Double-Blind, Vehicle-Controlled, PArallel Group Study of the Safety and Effectiveness of A-101 Solution 40% in Subjects With Seborrheic Keratosis on the Trunk, Extremities and Face.
Brief Title: A Randomized, Double-Blind, Vehicle-Controlled Study in Subjects With Seborrheic Keratosis
Acronym: SK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-101-SEBK-302
Record Dates: First submitted 2016-01-26; First posted 2016-01-28 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2016-01

CONDITIONS: Seborrheic Keratosis
Keywords: seborrheic keratosis
MeSH Terms: conditions — Keratosis, Seborrheic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A-101 Solution (Experimental): A-101 Solution 40% administered once
  Interventions: Drug: A-101 Solution
- Vehicle Solution (Placebo Comparator): Vehicle Solution administered once
  Interventions: Other: Vehicle Solution

INTERVENTIONS:
Drug: A-101 Solution
  Arms: A-101 Solution
Other: Vehicle Solution — Placebo
  Arms: Vehicle Solution

SUMMARY:
This is a randomized, double-blind, vehicle-controlled, parallel group study.

DETAILED DESCRIPTION:
This is a randomized, double-blind, vehicle-controlled, parallel group study. During this study, the investigator will identify 4 eligible SK Target Lesions on each subject on the trunk, extremities and face.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Clinical diagnosis of stable clinically typical seborrheic keratosis
3. Subject has 4 appropriate seborrheic keratosis Target Lesions on the trunk, extremities and face that each are eligible for treatment as defined below:

   * Have a clinically typical appearance
   * Have a PLA of 2 or greater and be a discrete lesion
   * Not be covered with hair which, in the investigator's opinion, would interfere with the study medication treatment or the study evaluations
   * Not be in an intertriginous fold
   * Not be on the eyelids
   * Not be within 5mm of the orbital rim
   * Not be pedunculated
4. If the subject is a woman of childbearing potential, she has a negative urine pregnancy test and agrees to use an active method of birth control for the duration of the study
5. Subject is non-pregnant and non-lactating
6. Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of any Target Lesion or which exposes the subject to an unacceptable risk by study participation
7. Subject is willing and able to follow all study instructions and to attend all study visits
8. Subject is able to comprehend and willing to sign an Informed Consent Form.

Exclusion Criteria:

1. Subject has clinically atypical and - or rapidly growing seborrheic keratosis lesions 2. Subject has presence of multiple eruptive seborrheic keratosis lesions (Sign of Lesser -Trelat) 3. Subject has a current systemic malignancy 4. Subject has used any of the following systemic therapies within the specified period prior to enrollment:

* Retinoids; 180 days
* Glucocortico-steroids;
* Anti-metabolites (e.g., methotrexate); 5. Subject has used any of the following topical therapies within the specified period or in a proximity to any Target Lesion, that in the investigator's opinion interferes with the study medication treatment or the study assessments:
* LASER, light or other energy based therapy (e.g., intense pulsed light, photo-dynamic therapy;
* Liquid nitrogen, electrodesiccation, curettage, imiquimod, 5-flurouracil, or ingenol mebutate;
* Retinoids;
* Microdermabrasion or superficial chemical peels;
* Glucocortico-steroids or antibiotics 6. Subject currently has or has had any of the following within the specified period or in a proximity to any Target Lesion that, in the investigator's opinion, interferes with the study medication treatment or the study assessments:
* A cutaneous malignancy;
* A sunburn; currently
* A pre-malignancy (e.g., actinic keratosis); currently
* Body art (e.g., tattoos, piercing, etc.); currently
* Excessive tan; currently 7. Subject has a history of sensitivity to any of the ingredients in the study medications 8. Subject has any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or condition (e.g., sunburn, excessive hair, open wounds) that, in the opinion of the investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations 9. Subject has participated in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Shanler, MD, Study Director — Aclaris Therapeutics, Inc.
Locations (1):
- Aclaris Therapeutics, Inc., Malvern, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smith SR, Xu S, Estes E, Shanler SD. Anatomic Site-Specific Treatment Response With 40% Hydrogen Peroxide (w/w) Topical Formulation for Raised Seborrheic Keratoses: Pooled Analysis of Data from Two Phase 3 Studies. J Drugs Dermatol. 2018 Oct 1;17(10):1092-1098. PMID 30365590

RESULTS

PARTICIPANT FLOW:
Groups:
- A-101 Solution: A-101 Solution 40% administered once
  A-101 Solution
Period: Overall Study
Arm/Group | A-101 Solution | Vehicle Solution
Started | 244 | 243
Completed | 233 | 228
Not Completed | 11 | 15
Not completed — Protocol Violation | 11 | 7
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Discontinued early without completing | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A-101 Solution | Vehicle Solution | Total
Number analyzed (Participants) | 244 | 243 | 487
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 74 | 156
  >=65 years | 162 | 169 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.92) | 69.1 (8.64) | 68.7 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 136 | 284
  Male | 96 | 107 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 26
  Not Hispanic or Latino | 229 | 222 | 451
  Unknown or Not Reported | 3 | 7 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 241 | 236 | 477
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 244 | 243 | 487

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With All Target Lesions Cleared According to Physician Lesion Assessment Scale
Description: Proportion of subjects for whom all target lesions were judged to be clear on the Physician Lesion Assessment Scale (PLA=0) at Visit 8. The Physician Lesion Assessment Scale is a 4 point scale used by the investigator to assess the subject's target sk lesions.
Time Frame: Study day 106
Measure: Count of Participants; unit: Participants
Arm/Group | A-101 Solution | Vehicle Solution
Number analyzed (Participants) | 244 | 243
Participants | 19 | 0

2. Secondary Outcome: Percent of Lesions Cleared Scale
Description: Proportion of Subjects for whom at least 3 of 4 target lesions were judged to be clear on the Physician Lesion Assessment Scale (PLA=0) at Visit 8
Time Frame: Study day 106
Measure: Count of Participants; unit: Participants
Arm/Group | A-101 Solution | Vehicle Solution
Number analyzed (Participants) | 244 | 243
Participants | 56 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from V2 (Day 1) through V8 (Day 106)
Arm/Group | A-101 Solution | Vehicle Solution
All-Cause Mortality (participants affected / at risk) | 0/244 | 0/243
Serious Adverse Events (participants affected / at risk) | 6/244 | 4/243
Other Adverse Events (participants affected / at risk) | 8/244 | 7/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-101 Solution (N=244) | Vehicle Solution (N=243)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Node Dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Pubis Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast Cancer Stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Precerebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Post traumatic Stress Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-101 Solution (N=244) | Vehicle Solution (N=243)
Sinusitis (Infections and infestations) | 4 (4) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3)
Herpes Zoster (Infections and infestations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and Investigator agree not to publish the results of this study without the prior written consent of the Sponsor.